CLINICAL TRIAL: NCT05117281
Title: Comparison of Postoperative Analgesic Efficacy of Caudal Block Versus Spinal Block With Levobupivacaine for Inguinal Hernia in Children: A Randomized Clinical Trial
Brief Title: Comparison of Postoperative Analgesic Efficacy of Caudal Block Versus Spinal Block With Levobupivacaine for Inguinal Hernia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17300727
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pain, Postoperative; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal group (Active Comparator): Plain, isobaric levobupivacaine(0.25%) 0.25 mg/kg
  Interventions: Drug: Levobupivacaine
- caudal group (Active Comparator): Plain, isobaric levobupivacaine (0.25%) 1 ml/kg
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Plain, isobaric levobupivacaine (0.25%) 1 ml/kg
  Other Names: Levobupivacaine hydrate
  Arms: caudal group
Drug: Levobupivacaine — Plain, isobaric levobupivacaine (0.25%) 0.25 mg/kg
  Other Names: levobupivacaine hydrate
  Arms: spinal group

SUMMARY:
Neuraxial analgesia may improve postoperative outcomes for high-risk children who are susceptible to respiratory complications (e.g. post-operative apnea). The use of spinal anesthesia in infants and children requiring surgeries of the sub-umbilical regions is gaining considerable popularity worldwide. Caudal analgesia along with general anesthesia is a very popular regional technique for prolonged postoperative analgesia in different pediatric surgical procedures where the surgical site is sub-umbilical. Bupivacaine has been thoroughly studied, and a large global experience exists.

DETAILED DESCRIPTION:
Neuraxial analgesia may improve postoperative outcomes for high-risk children who are susceptible to respiratory complications (post-operative apnea). In this population, spinal anesthesia has been proposed as a means to reduce post-operative complications, especially apnea and post-operative respiratory dysfunction, although this utility has been questioned.

Spinal anesthesia modifies the neuroendocrine stress response, ensures a more rapid recovery, and may shorten hospital stay with fewer opioid-induced side effects.

Caudal analgesia along with general anesthesia is a very popular regional technique for prolonged postoperative analgesia in different pediatric surgical procedures where the surgical site is sub-umbilical. Caudal anesthetics usually provide an-algesia for approximately 4-6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-10 years.
* Weight: 15-40 kg.
* Sex: both males and females.
* ASA physical status: 1-II.
* Operation: surgery below the umbilicus.

Exclusion Criteria:

* Allergic reaction to local anesthetics (LAs).
* Local or systemic infection (risk of meningitis).
* Intracranial hypertension.
* Hydrocephalus.
* Intracranial hemorrhage.
* Coagulopathy.
* Hypovolemia.
* Parental refusal.
* Spinal deformities, such as spina bifida or myelomeningocele.
* Presence of a ventriculoperitoneal shunt because of a risk of shunt infection or dural leak.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
FLACC scale FLACC scores will be recorded. FLACC scores will be recorded. FLACC score will be recorded | 24 hours postoperative
  Face, Legs, Activity, Cry, Consolability scale will be recorded. Each category is scored on the 0 to 2 scale. Add the scores together (for a total possible score of 0 to 10).

SECONDARY OUTCOMES:
Total consumption of rescue analgesics | 24 hours
  mg/24

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt